CLINICAL TRIAL: NCT06077240
Title: Evaluating The Effects Of E-cigarettes Versus Oral Nicotine Pouches and Product Constituents (Menthol Flavor, Nicotine Concentration) On Adult Cigarette Smoking and Addiction
Brief Title: Effects of E-cigs vs Pouches on Cigarette Smoking and Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000035286; U54DA036151 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Smoking; Smoking Behaviors; Nicotine Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems; Nicotine; Menthol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To avoid randomized non-starters and potential bias due to differential early attrition from prior knowledge of group assignment, randomization will occur at the time of visit 0 when participants first receive tobacco products specific to their assigned condition, and neither the research assistant nor participant will know the assignment in advance. Researchers and participants will be blinded to the nicotine concentration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarettes (Experimental): Adults who smoke cigarettes will be randomized to receive e-cigarettes for a duration of 4 weeks and to 1 of 4 possible regulatory scenarios within products where flavor availability is either menthol and tobacco/unflavored available or tobacco/unflavored only available, and nicotine concentration is either higher (5% e-cig) or lower (2.4% e-cig). Participants will return for bi-weekly research visits (in person or remote videocall) to complete measures for study aims. They will complete a final follow-up at Week 6 to assess maintenance of cigarette reduction and willingness to continue using products once they are no longer provided.
  Interventions: Behavioral: E-cigarette with 2.4% Nicotine with Menthol and Tobacco Flavors; Behavioral: E-cigarette with 2.4% Nicotine with Tobacco Flavor Only; Behavioral: E-cigarette with 5% Nicotine with Menthol and Tobacco Flavors; Behavioral: E-cigarette with 5% Nicotine with Tobacco Flavor Only
- Nicotine Pouches (Experimental): Adults who smoke cigarettes will be randomized to receive nicotine pouches for a duration of 4 weeks and to 1 of 4 possible regulatory scenarios within products where flavor availability is either menthol and tobacco/unflavored available or tobacco/unflavored only available, and nicotine concentration is either higher (6mg pouch) or lower (3mg pouch). Participants will return for bi-weekly research visits (in person or remote videocall) to complete measures for study aims. They will complete a final follow-up at Week 6 to assess maintenance of cigarette reduction and willingness to continue using products once they are no longer provided.
  Interventions: Behavioral: Tobacco Pouches with 3mg Nicotine with Menthol and Tobacco Flavors; Behavioral: Tobacco Pouches with 3mg Nicotine with Tobacco Flavor Only; Behavioral: Tobacco Pouches with 6mg Nicotine with Menthol and Tobacco Flavors; Behavioral: Tobacco Pouches with 6mg Nicotine with Tobacco Flavor Only

INTERVENTIONS:
Behavioral: E-cigarette with 2.4% Nicotine with Menthol and Tobacco Flavors — Flavor availability is menthol and tobacco/unflavored with lower nicotine concentration.
  Arms: E-cigarettes
Behavioral: E-cigarette with 2.4% Nicotine with Tobacco Flavor Only — Flavor availability is tobacco/unflavored only with lower nicotine concentration.
  Arms: E-cigarettes
Behavioral: E-cigarette with 5% Nicotine with Menthol and Tobacco Flavors — Flavor availability is menthol and tobacco/unflavored with higher nicotine concentration.
  Arms: E-cigarettes
Behavioral: E-cigarette with 5% Nicotine with Tobacco Flavor Only — Flavor availability is tobacco/unflavored only with higher nicotine concentration.
  Arms: E-cigarettes
Behavioral: Tobacco Pouches with 3mg Nicotine with Menthol and Tobacco Flavors — Flavor availability is menthol and tobacco/unflavored with lower nicotine concentration.
  Arms: Nicotine Pouches
Behavioral: Tobacco Pouches with 3mg Nicotine with Tobacco Flavor Only — Flavor availability is tobacco/unflavored only with lower nicotine concentration.
  Arms: Nicotine Pouches
Behavioral: Tobacco Pouches with 6mg Nicotine with Menthol and Tobacco Flavors — Flavor availability is menthol and tobacco/unflavored with higher nicotine concentration.
  Arms: Nicotine Pouches
Behavioral: Tobacco Pouches with 6mg Nicotine with Tobacco Flavor Only — Flavor availability is tobacco/unflavored only with higher nicotine concentration.
  Arms: Nicotine Pouches

SUMMARY:
The study will recruit an anticipated 256 adults who currently smoke cigarettes and report a willingness to try switching to alternative, non-combustible products. Participants will be randomized to receive either e-cigarettes or nicotine pouches for a duration of 4 weeks and to 1 of 4 possible regulatory scenarios within products where flavor availability is either menthol and tobacco/unflavored available or tobacco/unflavored only available, and nicotine concentration is either higher (5% e-cig, 6mg pouch) or lower (2.4% e-cig, 3mg pouch). Participants will return for bi-weekly research visits (in person or remote videocall) to complete measures for study aims. Participants will complete a final follow-up at Week 6 to assess maintenance of cigarette reduction and willingness to continue using products once they are no longer provided. The investigators expect to observe which products and constituents lead to greater smoking reduction.

DETAILED DESCRIPTION:
The study includes 5 visit and assessments over 6 weeks. The intake visit will take approximately 60 minutes and subsequent visits will take approximately 30 minutes. The study is proposed to run for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years old
* English literate
* Currently smoking cigarettes, biochemically confirmed
* Not planning a smoking cessation attempt or to use smoking cessation pharmacotherapies (NRT, bupropion, varenicline) in the next month.

Exclusion Criteria:

* Currently using any smoking cessation services and/or pharmacotherapies
* Currently pregnant or breastfeeding
* Significant current medical or psychiatric condition
* Known hypersensitivity to propylene glycol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Average number of cigarettes smoked per day | From baseline to week 4
  Participants will report the total number of cigarettes consumed each day using a well-validated timeline follow-back (TLFB) interview method to assess number of cigarettes smoked per day continuously over the 4-week observational period for each product condition.
Aim 2: Percent of days using non-combustible product | From baseline to week 4
  Participants will report daily use of e-cigarettes or nicotine pouches using a well-validated timeline follow-back (TLFB) interview method continuously over the 4-week observational period to determine the total percent days use of the non-combustible product for each product condition.

SECONDARY OUTCOMES:
Aim 1: Percent of days abstinent from cigarettes | From baseline to week 4
  Participants will report the total number of cigarettes consumed each day using a well-validated timeline follow-back (TLFB) interview method to assess number of cigarettes smoked per day continuously over the 4-week observational period to determine the total percent days abstinent (smoke-free) for each product condition.
Aim 1: Biochemically verified 7 day point-prevalent abstinence from cigarettes | Week 4
  Complete switching from cigarettes will be assessed at the end of the study period using self-reported TLFB methods and biochemical verification with expired breath carbon monoxide (CO) testing (CO < 5ppm) to determine rates of 7-day point-prevalent abstinence
Aim 1: Cigarette Dependence | From baseline to week 4
  Cigarette dependence will be measured using the 4-item PROMIS® Short Form v1.0 - Smoking Nicotine Dependence for All Smokers 4a. Each item is scored from 1-5 with the range of scores from 4-20 with higher scores representing greater cigarette dependence.
Aim 2: Average use of non-combustible products per day | From baseline to week 4
  Participants will report daily e-cigarette and nicotine pouch quantity and frequency consumed using a well-validated timeline follow-back (TLFB) interview method to use continuously over the 4-week observational period for each product condition.
Aim 2: Continued use of non-combustible products | Week 4 to 6
  Participants will report daily use of e-cigarettes or nicotine pouches using a well-validated timeline follow-back (TLFB) interview method to determine the total percent days use of the non-combustible product for each product condition during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, PhD, Principal Investigator — Yale University; Krysten Bold, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available through the NIH repository- National Addiction & HIV Data Archive Program (NAHDAP)
Time Frame: After study completion
Access Criteria: Available upon request